CLINICAL TRIAL: NCT05341427
Title: DEVELOPMENT OF A CLINICAL PREDICTION RULES TO IDENTIFY EFFICACY OF PULSED ELECTROMAGNETIC THERAPY ON BURN WOUND HEALING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed mohamed nagy, lecturer of physical therapy for surgery- cairo university, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003534
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Burn Wound
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- burn wound receiving electromagnetic therapy (Experimental): There will be only one intervention group. The duration of the study will be 6 weeks divided to 18 sessions (three sessions per week). Sixty patients (male and female) will be recruited from the burn units of Cairo university hospitals
  Interventions: Device: electromagnetic device

INTERVENTIONS:
Device: electromagnetic device — electromagnetic waves for burn wound

SUMMARY:
The purpose of this study is to investigate whether patients' age, total burned surface area, wound stage and wound depth determine wound healing response to pulsed electromagnetic therapy in burn patients

DETAILED DESCRIPTION:
It will be hypothesized that

1. Age may significantly affect burn wound healing's response to pulsed electromagnetic waves.
2. TBSA may significantly affect burn wound healing's response to pulsed electromagnetic waves
3. Depth of wound may significantly affect burn wound healing's response to pulsed electromagnetic waves
4. Wound healing stage may significantly affect burn wound healing's response to pulsed electromagnetic waves This study will be conducted at the in-patient burn units. There will be only one intervention group. The duration of the study will be 6 weeks divided to 18 sessions (three sessions per week). Sixty patients (male and female) will be recruited from the burn units.

Pulsed electromagnetic waves will be performed for 60 min 3 times per week till healing (maximum 8 weeks) on the wound area.

PEMF therapy will be as (duration: 60 minutes; frequency: 12 Hz; intensity: 12 Gauss)

ELIGIBILITY:
Inclusion Criteria Partial thickness Burn wound depth. Age ranges from 20-50 years. TBSA more than 15% Sufficient understanding to perform the tests. Exclusion Criteria Diabetic patients. Patients receiving immunosuppressive drugs. Associated co-morbidities, such as neurological diseases, malnutrition, and other inﬂammatory and/or infectious diseases.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
wound healing rate | maximum of 6 weeks
  tools for assessment of wound area changes before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No